CLINICAL TRIAL: NCT00620451
Title: A Phase IIb, Randomized, Double-Blind, Placebo Controlled Study for the Treatment of Active Celiac Disease With Larazotide Acetate (AT-1001)
Brief Title: Randomized, Double-Blind, Placebo-Controlled Study of Larazotide Acetate in Subjects With Active Celiac Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 9 Meters Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AT1001-011
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Celiac Disease
Keywords: Treatment; Active; Celiac; Remission; Induction
MeSH Terms: conditions — Celiac Disease; Motor Activity | interventions — larazotide acetate

STUDY DESIGN:
Intervention Model Description: randomized, parallel- group, double-blind, multicenter
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Larazotide acetate 4 mg (Experimental): larazotide acetate capsules 4 mg TID
  Interventions: Drug: larazotide acetate
- Larazotide acetate 8 mg (Experimental): Larazotide acetate capsules 8 mg TID
  Interventions: Drug: larazotide acetate
- Placebo (Placebo Comparator): Placebo capsules
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: larazotide acetate — gelatin capsule
  Other Names: AT-1001; INN-202
  Arms: Larazotide acetate 4 mg; Larazotide acetate 8 mg
Drug: placebo — gelatin capsule
  Arms: Placebo

SUMMARY:
This study was conducted to assess the safety and efficacy of larazotide acetate versus placebo in inducing remission in subjects with active celiac disease.

DETAILED DESCRIPTION:
This was an outpatient, randomized, parallel- group, double-blind, multicenter, 8-week study with three treatment arms: larazotide acetate 4 mg TID, larazotide acetate 8 mg TID and placebo TID in subjects with celiac disease. The primary objective was to assess the efficacy of larazotide acetate versus placebo in inducing remission in subjects with active celiac disease, as defined by an improvement in the Villous Height to Crypt Depth (Vh:Cd) ratio, obtained by duodeno-jejunal biopsy. Secondary objectives included assessment of the safety and tolerability of larazotide acetate, to prospectively validate the components of a composite weighted index of celiac disease activity (celiac disease Activity Rating Score, CeDARS), individually and as a whole, to To compare the CeDARS against the Clinician Global Assessment of disease (CGA), Psychological Well Being Index and the Short Form 12 version 2 (SF-12 v2) health survey and to assess the effects of larazotide acetate on inflammatory markers in subjects with active celiac disease.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults with celiac disease (as demonstrated by duodenal/jejunal biopsy or by capsule endoscopy plus positive anti-tTG)
* Marsh score ≥ II at screening
* Positive serum anti-tTG antibodies as determined by screening serology
* Willing to comply with a gluten-free diet for the duration of the study

Exclusion Criteria:

* Has refractory Celiac Disease or severe complications of celiac disease (eg, EATL-, ulcerative jejunitis, perforation, etc.)
* Has chronic active GI disease other than Celiac Disease
* Has diabetes (Type 1 or Type 2) or other autoimmune disease that might interfere with the conduct of the study
* Has hemoglobin value below 8.5 g/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Assess the efficacy of larazotide acetate in inducing remission in subjects with active celiac disease | duodeno-jejunal biopsies were performed at Baseline and Day 56
  Remission was defined as an improvement in the Villous Height to Crypt Depth (Vh:Cd) ratio obtained by duodeno-jejunal biopsy.

SECONDARY OUTCOMES:
Assess the safety and tolerability of larazotide acetate | Up to 8 weeks
  Safety endpoints assessed in this study were adverse events, vital signs, physical examination results, clinical laboratory test results and ECG results. Plasma larazotide acetate and metabolites, as well as potential serum antibodies against larazotide acetate, were also determined.
To prospectively validate the components of a composite weighted index of Celiac Disease activity (Celiac Disease Activity Rating Score, CeDARS), individually and as a whole. | Up to 8 weeks
  Candidate components of the CeDARS Index measured in this study were GSRS, anti-tTG antibodies, LAMA ratio, Hb, ferritin, body weight, triceps skin fold thickness, BMI, urinary nitrates
To compare the CeDARS against the Clinician Global Assessment of disease (CGA), Psychological Well Being Index (PWBI) and the Short Form 12 version 2 (SF-12v2) health survey. | CGA, PWBI and SF-12v2 were collected at Visits 2, 3 and 4.
  The CGA was completed by the PI or designee; the PWBI and SF-12v2 were completed by the subject.
To assess the effects of larazotide acetate on inflammatory markers in subjects with active celiac disease subjects | Blood draws occurred at Visits 1, 2, 3, 4 and 5.
  Blood for serum was drawn for potential future determination of inflammatory mediators that might be involved in the response of Celiac Disease to larazotide acetate, such as cytokines (e.g. TNF-α,IFN-γ) or the putative permeability factor "zonulin".

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Leon, MD, Ph.D, Study Director — Alba Therapeutics
Locations (32):
- United States (20):
  - Study Site, Orange, California
  - Study Site, San Francisco, California
  - Study Site, Torrington, Connecticut
  - Study Site, Jacksonville, Florida
  - Study Site, Topeka, Kansas
  - Study Site, Lexington, Kentucky
  - Study Site, Hagerstown, Maryland
  - Study Site, Silver Spring, Maryland
  - Study Site, Chesterfield, Michigan
  - Study Site, Troy, Michigan
  - Study Site, Rochester, Minnesota
  - Study Site, Asheville, North Carolina
  - Study Site, Harrisburg, North Carolina
  - Study Site, Gallipolis, Ohio
  - Study Site, Paoli, Pennsylvania
  - Study Site, Philadelphia, Pennsylvania
  - Study Site, Pittsburgh, Pennsylvania
  - Study Site, Sioux Falls, South Dakota
  - Study Site, Franklin, Tennessee
  - Study Site, Houston, Texas
- Canada (4):
  - Study Site, Edmonton, Alberta
  - Study Site, Abbotsford, British Columbia
  - Study Site, Kelowna, British Columbia
  - Study Site, Richmond Hill, Ontario
- Spain (8):
  - Study Site, Palma, Mallorca
  - Study Site, Barcelona
  - Study Site, Huesca
  - Study Site, León
  - Study Site, Madrid
  - Study site, Madrid
  - Study Site, Reus
  - Study Site, Valladolid